CLINICAL TRIAL: NCT04877431
Title: Post Authorization Study to Monitor Efficacy, Effectiveness and Safety of Teduglutide (Revestive®) in Adult and Pediatric Patients With Short Bowel Syndrome in Argentina
Brief Title: A Study of Teduglutide (Revestive®) in Children, Teenagers and Adults With Short Bowel Disease
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-633-4003
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- De Nova Participants: De nova participants who had received teduglutide after marketing authorization will be enrolled in this study and monitored by their physicians according to local clinical practice then followed for 24-weeks unless treatment discontinuation or lost to follow-up.
- Legacy Participants: Legacy participants who received teduglutide treatment prior to marketing authorization under expanded access type of program will be enrolled in this study and monitored by their physicians according to local clinical practice then followed for 24-weeks unless treatment discontinuation or lost to follow-up.

SUMMARY:
The main aims of the study are to assess the safety profile of Teduglutide (Revestive®) in people with Short Bowel Disease as well as how well people respond to the treatment with Teduglutide (Revestive®).

This study is about collecting data only; participants receive Teduglutide (Revestive®) by their doctors according to the clinical practice but not as part of this study. Only standard care information available in the participant's medical records will be reviewed and collected for this study.

Participants do not need to visit their doctor in addition to their normal visits.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants (greater than or equal to [>=] 18 years) or pediatric (>= 1 year and less than [<] 18) with a diagnosis of SBS who are dependent on parenteral support.
* Have received at least one dose of teduglutide according to approved indications.
* Signed the mandatory consent that has been agreed with national regulatory authorities (ANMAT) as applicable.

Exclusion Criteria:

- Not Applicable.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All adult and pediatric participants who are treated with teduglutide according to approved indications.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events of Special Interest (AESI) | Up to 24 months
  AESI will include biliary disorders and cholecystitis; pancreatic disease; cardiovascular adverse events associated with fluid overload; intestinal obstruction; stoma complications; malignancy; gastrointestinal neoplastic growth, including colorectal polys and small bowel neoplasia; adverse events associated with increased absorption of concomitant oral medications; anxiety; injection site reactions and suspected immunogenic reactions (like hypersensitivity or other reactions); embryo-fetal toxicity (assessed through follow up of all pregnancies).
Number of Participants With Adverse Events (AEs) | Up to 24 months
  An AE is any untoward medical occurrence in a participant administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment. A serious adverse events (SAEs) is any untoward clinical manifestation of signs, symptoms or outcomes (whether considered related to investigational product or not and at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of hospitalization, results in persistent or significant disability/incapacity, congenital abnormality/birth defect, an important medical event. Number of participants with AEs including serious and non-serious AEs will be assessed.

SECONDARY OUTCOMES:
Percentage of Participants With Clinical Response at Week 12 and 24 | Week 12 and 24
  Clinical response will be defined as a 20 percent (%) or more reductions on weekly parenteral support volume.
Change From Baseline in Weekly Parenteral Support Volume at Week 12 and 24 | Baseline, Week 12 and 24
  Parenteral support volume will be assessed at baseline (before treatment), and at Week 12, and 24.
Change From Baseline in Number of Days per Week of Parenteral Support at Week 12 and 24 | Baseline, Week 12 and 24
  Change from baseline in number of days per week requiring parenteral support will be assessed at baseline (before treatment), and at Week 12 and 24.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- IC Projects, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/60990714ef0b71001e743c57